CLINICAL TRIAL: NCT04801173
Title: Effect of Very Low Calorie Ketogenic Diet on Obese and Insulin-resistant Women With Polycystic Ovary Syndrome: a Controlled Randomized Trial
Brief Title: Ketogenic Diet in PCOS With Obesity and Insulin Resistance
Acronym: VLCKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Pronokal group (Unknown)
Responsible Party: Principal Investigator, Alessandra Gambineri, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLCKD
Record Dates: First submitted 2021-03-01; First posted 2021-03-16 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: PCOS; Obesity; Insulin Resistance
Keywords: Ketogenic diet; Insulin resistance; PCOS; Obesity; Hyperandrogenism
MeSH Terms: conditions — Obesity; Insulin Resistance; Hyperandrogenism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very low calorie ketogenic diet (Experimental): Dietary intervention with a very low calorie ketogenic diet, using commercial products of the Pronokal PnK® method
  Interventions: Combination Product: Very low calorie ketogenic diet; Behavioral: Low calorie standard diet
- Low calorie diet (Active Comparator): Control treatment with a low calorie standard diet
  Interventions: Behavioral: Low calorie standard diet

INTERVENTIONS:
Combination Product: Very low calorie ketogenic diet — Dietary intervention with a very low calorie ketogenic diet, using commercial products of the Pronokal PnK® method
  Other Names: Pronokal method
  Arms: Very low calorie ketogenic diet
Behavioral: Low calorie standard diet — Low calorie standard diet with no specified dietary supplement addition

SUMMARY:
The purpose of the VLCKD randomized clinical trial is to demonstrate the superiority of very low calorie ketogenic diet with respect to the standard low calorie diet in reducing body weight and insulin resistance in obese and insulin resistant patients with Polycystic Ovary Syndrome

DETAILED DESCRIPTION:
Consecutive patients coming to the Endocrinology and Diabetes Clinic of the S.Orsola hospital in Bologna with the suspicion of PCOS, during the study period, will be eligible to participate. In the screening phase, patients from the clinic conforming to the inclusion criteria will be invited to participate in the anovulation screening phase, lasting up to 8 weeks, during which measurements of LH, FSH, estradiol, progesterone and a gynecologic ultrasound will be done on 7th, 14th, 21st and 28th day of the presumed ovulatory cycle, or at any time if amenorrhea present. Consenting participants will provide written informed consent.

Following the anovulation screening, the patients will be randomized in two arms of the study: 1. very low calorie ketogenic diet (VLCKD) and the 2. low calorie standard diet (LCD).

The study is open label; thus, patients and investigators will not be blinded to treatment allocation due to the nature of the study intervention.

The group assigned to the VLCKD will follow the VLCKD for 8 weeks, after which they will follow the LCD for the next 8 weeks.

The group assigned to the LCD will follow the LCD for the entire length of the study (16 weeks.)

At the start of the study, after 8 weeks and after 16 weeks, following measurements and tests will be done:

1. clinical examination with the measurement of height, body mass, circumference at the waist and hip level, arterial systolic and diastolic pressure, heart rate, Ferriman-Gallwey and videodermoscopic evaluation of hirsutism and bioimpedance body composition measurement;
2. blood will be taken for: lipid profile, hepatic transaminases, fasting glucose, fasting insulin, HbA1c, potassium, sodium, urea, calcium, phosphorus, total proteins, albumins, total bilirubin, uric acid, complete blood count, sex hormone binding globulin (SHBG), liquid chromatography-mass spectrometry measurement of testosterone, androstenedione, DHEA, 17OH-progesterone, 17OH-pregnenolone;
3. dietary interview;
4. psychological evaluation using the following questionnaires: Symptom Questionnaire, the Psychosocial index and the Psychological Well-Being scales.

ELIGIBILITY:
Inclusion Criteria:

* PCOS according to the NIH criteria;
* Body mass index (BMI) between 30 and 35 kg/m3;
* HOMA index ≥ 3 (according to formula: (fasting glucose [mmol/L] × fasting insulin [mIU/L])/22.5)
* Written informed consent.

Exclusion Criteria:

* Diabetes type 1
* Exogenous insulin or insulin analogue therapy
* Obesity caused by endocrine disease other than PCOS
* Obesity caused by pharmacotherapy
* Use of a weight-loss diet in the past 3 months
* Use of contraceptive pills in the past 3 months
* Severe depression
* Other psychiatric diseases
* Alcohol or psychoactive substance abuse
* Severe hepatic insufficiency
* Renal calculosis
* Renal insufficiency
* Episodes of gout
* Malignant neoplasia
* Previous cardiovascular or cerebrovascular events
* Uncontrolled hypertension
* Water-electrolyte imbalance
* Any pharmacotherapy capable of interfering with glucose metabolism
* Any pharmacotherapy capable of interfering with steroid metabolism
* Menopause
* Pregnancy
* Lactation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Body mass index | 16 weeks after the start of treatment
  Weight and height will be combined to report BMI in kg/m^2
Change in body composition measured by bioimpedentiometry | 16 weeks after the start of the treatment
  Fat mass and lean mass changes will be considered to estimate change in body composition and reported as %

SECONDARY OUTCOMES:
Change in Body mass index | 8 weeks after the start of treatment
  Weight and height will be combined to report BMI in kg/m^2
Change in body composition measured by bioimpedentiometry | 8 weeks after the start of the treatment
  Fat mass and lean mass will be considered to estimate change in body composition and reported as %
Change in Homeostasis Model Assessment Index | 16 weeks after the start of the treatment
  Fasting glucose in mmol/L and fasting insulin in mcU/mL will be combined to report Homeostasis Model Assessment Index
Change in frequency of menstrual cycles | 16 weeks after the start of the treatment
  Number of menses in the 16 weeks before will be considered to report the frequency of menstrual cycles
Change in hirsutism | 16 weeks after the start of the treatment
  Modified Ferriman-Gallwey score will be used to measure changes in hirsutism; the minimum and maximum values are 4 and 36 respectively; higher score means a worse outcome
Change in plasma concentrations of testosterone | 16 weeks after the start of the treatment
  testosterone will be reported in ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Endocrinology and Prevention and Care of Diabetes, S.Orsola Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tosi F, Bonora E, Moghetti P. Insulin resistance in a large cohort of women with polycystic ovary syndrome: a comparison between euglycaemic-hyperinsulinaemic clamp and surrogate indexes. Hum Reprod. 2017 Dec 1;32(12):2515-2521. doi: 10.1093/humrep/dex308. PMID 29040529
- [Background] Conway G, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Franks S, Gambineri A, Kelestimur F, Macut D, Micic D, Pasquali R, Pfeifer M, Pignatelli D, Pugeat M, Yildiz BO; ESE PCOS Special Interest Group. The polycystic ovary syndrome: a position statement from the European Society of Endocrinology. Eur J Endocrinol. 2014 Oct;171(4):P1-29. doi: 10.1530/EJE-14-0253. Epub 2014 May 21. PMID 24849517
- [Background] Repaci A, Gambineri A, Pasquali R. The role of low-grade inflammation in the polycystic ovary syndrome. Mol Cell Endocrinol. 2011 Mar 15;335(1):30-41. doi: 10.1016/j.mce.2010.08.002. Epub 2010 Aug 11. PMID 20708064
- [Background] Barrea L, Marzullo P, Muscogiuri G, Di Somma C, Scacchi M, Orio F, Aimaretti G, Colao A, Savastano S. Source and amount of carbohydrate in the diet and inflammation in women with polycystic ovary syndrome. Nutr Res Rev. 2018 Dec;31(2):291-301. doi: 10.1017/S0954422418000136. Epub 2018 Jul 23. PMID 30033891
- [Background] Gonzalez F. Nutrient-Induced Inflammation in Polycystic Ovary Syndrome: Role in the Development of Metabolic Aberration and Ovarian Dysfunction. Semin Reprod Med. 2015 Jul;33(4):276-86. doi: 10.1055/s-0035-1554918. Epub 2015 Jul 1. PMID 26132932
- [Background] Volk KM, Pogrebna VV, Roberts JA, Zachry JE, Blythe SN, Toporikova N. High-Fat, High-Sugar Diet Disrupts the Preovulatory Hormone Surge and Induces Cystic Ovaries in Cycling Female Rats. J Endocr Soc. 2017 Nov 2;1(12):1488-1505. doi: 10.1210/js.2017-00305. eCollection 2017 Dec 1. PMID 29308444
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Matsuzaki T, Douchi T, Oki T, Ishihara O, Okagaki R, Kajihara T, Tamura M, Kotsuji F, Tajima K, Kawano M, Ishizuka B, Irahara M. Weight reduction using a formula diet recovers menstruation in obese patients with an ovulatory disorder. Reprod Med Biol. 2017 Jul 7;16(3):268-275. doi: 10.1002/rmb2.12034. eCollection 2017 Jul. PMID 29259477
- [Background] Mehrabani HH, Salehpour S, Amiri Z, Farahani SJ, Meyer BJ, Tahbaz F. Beneficial effects of a high-protein, low-glycemic-load hypocaloric diet in overweight and obese women with polycystic ovary syndrome: a randomized controlled intervention study. J Am Coll Nutr. 2012 Apr;31(2):117-25. doi: 10.1080/07315724.2012.10720017. PMID 22855917
- [Background] Gower BA, Goss AM. A lower-carbohydrate, higher-fat diet reduces abdominal and intermuscular fat and increases insulin sensitivity in adults at risk of type 2 diabetes. J Nutr. 2015 Jan;145(1):177S-83S. doi: 10.3945/jn.114.195065. Epub 2014 Dec 3. PMID 25527677
- [Background] Mavropoulos JC, Yancy WS, Hepburn J, Westman EC. The effects of a low-carbohydrate, ketogenic diet on the polycystic ovary syndrome: a pilot study. Nutr Metab (Lond). 2005 Dec 16;2:35. doi: 10.1186/1743-7075-2-35. PMID 16359551
- [Background] Caprio M, Infante M, Moriconi E, Armani A, Fabbri A, Mantovani G, Mariani S, Lubrano C, Poggiogalle E, Migliaccio S, Donini LM, Basciani S, Cignarelli A, Conte E, Ceccarini G, Bogazzi F, Cimino L, Condorelli RA, La Vignera S, Calogero AE, Gambineri A, Vignozzi L, Prodam F, Aimaretti G, Linsalata G, Buralli S, Monzani F, Aversa A, Vettor R, Santini F, Vitti P, Gnessi L, Pagotto U, Giorgino F, Colao A, Lenzi A; Cardiovascular Endocrinology Club of the Italian Society of Endocrinology. Very-low-calorie ketogenic diet (VLCKD) in the management of metabolic diseases: systematic review and consensus statement from the Italian Society of Endocrinology (SIE). J Endocrinol Invest. 2019 Nov;42(11):1365-1386. doi: 10.1007/s40618-019-01061-2. Epub 2019 May 20. PMID 31111407
- [Background] Costello MF, Misso ML, Balen A, Boyle J, Devoto L, Garad RM, Hart R, Johnson L, Jordan C, Legro RS, Norman RJ, Mocanu E, Qiao J, Rodgers RJ, Rombauts L, Tassone EC, Thangaratinam S, Vanky E, Teede HJ; International PCOS Network. Evidence summaries and recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome: assessment and treatment of infertility. Hum Reprod Open. 2019 Jan 4;2019(1):hoy021. doi: 10.1093/hropen/hoy021. eCollection 2019. PMID 31486807
- [Background] Moreno B, Bellido D, Sajoux I, Goday A, Saavedra D, Crujeiras AB, Casanueva FF. Comparison of a very low-calorie-ketogenic diet with a standard low-calorie diet in the treatment of obesity. Endocrine. 2014 Dec;47(3):793-805. doi: 10.1007/s12020-014-0192-3. Epub 2014 Mar 4. PMID 24584583
- [Background] Goday A, Bellido D, Sajoux I, Crujeiras AB, Burguera B, Garcia-Luna PP, Oleaga A, Moreno B, Casanueva FF. Short-term safety, tolerability and efficacy of a very low-calorie-ketogenic diet interventional weight loss program versus hypocaloric diet in patients with type 2 diabetes mellitus. Nutr Diabetes. 2016 Sep 19;6(9):e230. doi: 10.1038/nutd.2016.36. PMID 27643725